CLINICAL TRIAL: NCT03142217
Title: Characterization of the Profile of Dysarthria in Huntington's Disease, Using the Clinical Evaluation Battery of Dysarthria
Acronym: Huntington
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decision of investigator
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0005
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Dysarthria; Huntington Disease
MeSH Terms: conditions — Dysarthria; Huntington Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Huntington's Disease (Other)
  Interventions: Other: Study of dysarthria in patients with Huntington's disease

INTERVENTIONS:
Other: Study of dysarthria in patients with Huntington's disease — Study of dysarthria in patients with Huntington's disease

SUMMARY:
Huntington's disease is a hereditary disease of rare autosomal dominant transmission, both neurodegenerative and neuro-psychiatric. Clinically, there are motor symptoms (chorea), cognitive disorders (dementia) and psychiatric disorders.

Among motor disorders, dysarthria is a commonly found symptom. This is classically referred to as hyperkinetic dysarthria according to the criteria of Darley's classification. However, this old classification (1969) is only based on perceptual analysis and lack of specificity.

Moreover, in the course of the disease, chorea (control of the striatal attack D2) decreases to give place to a parkinsonian syndrome (control of the striatal attack D1) and the dysarthria also evolves towards a hypokinetic form . It also seems likely that cerebellar involvement (responsible for ataxia) contributes to dysarthria.

No studies have been published to date to characterize dysarthria in Huntington's disease in a quantified, objective and specific manner. However, Canan Ozsancak describes choreic dysarthria as heterogeneous according to the patients and variable according to the productions. A perceptual study reports an imprecision of the consonants, a lengthening of the pauses, a variable flow, an absence of modulation of the pitch and a hoarse voice.

Finally, few patients are cared for in speech therapy and there is no specific rehabilitation strategy: this would require - and justify a more precise study of the dysarthria of these patients.

The Clinical Evaluation of Dysarthria developed by Pascal Auzou and Véronique Rolland-Monnoury is a recent and partially standardized tool, combining qualitative and quantitative evaluation, which seems adapted to try to better characterize the dysarthria in Huntington's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Patients HD
* Major Patients
* French-speaking patients
* MMS score greater than 20
* Patients with informed consent signed
* Patients covered by a social insurance system

Exclusion Criteria:

* Patients with intercurrent pathologies or other psychiatric disorders that may interfere with battery replacement (at the discretion of the investigator)
* Illiteracy
* Persons placed under safeguard of justice (adults under guardianship or guardianship) or deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Analysis of the Clinical Evaluation Battery of Dysarthria using criteria to establish a clinical profile specific to Huntington's disease | 1 day